CLINICAL TRIAL: NCT00301314
Title: A Retrospective Study of Toxicity and Outcome of High Dose Chemotherapy With Autologous Stem Cell Transplant in Patients With Hodgkin Lymphoma (HL).
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Other Study IDs: 2655
Record Dates: First submitted 2006-03-09; First posted 2006-03-10 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Autologous stem cell transplant

SUMMARY:
The majority of patients with Hodgkin Lymphoma (HL)are cured with radiation therapy and/or combination chemotherapy. However, patients who relapse after attaining a complete remission with chemotherapy and those with primary refractory disease have a poor outcome with conventional chemotherapy regimens. Treatment results with standard-dose second-line regimens produce low complete remission rates and minimal survival benefit. Single institution studies have shown better outcome after autologous stem cell transplant in this group of patients when compared to historical controls receiving conventional treatment. In this retrospective review, we aim to analyze outcome and determine independent prognostic factors which would correlate with the long-term outcome of patients with HL who received an autologous stem cell transplant in the past at the Royal Marsden Hospital Eligible patients (those on current-follow-up) identified from the transplant database will be eligible for the study.

Accrual of eligible patients currently under follow-up will be performed in clinic at the time of next appointment. All patients accrued will give informed consent to participate in the study for retrospective case note review, after discussion with a study investigator and after receiving a study information sheet. The results of the analysis will be published in a peer-reviewed medical journal.

ELIGIBILITY:
Inclusion Criteria:

* a) Age over 18 b) Patients with Hodgkin Lymphoma who have received an autologous stem cell transplant c) Informed written consent

Exclusion Criteria:

* a) Medical or psychiatric conditions that compromise the patient's ability to give informed consent b) HIV positive or AIDS related lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 219 participants aged over 18 with Hodgkin Lymphina who have received an autologous stem cell transplant and written informed consent.
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, FRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS trust, Sutton, Surrey, United Kingdom